CLINICAL TRIAL: NCT01835665
Title: An Open Label Dose Finding Study of Nimodipine for the Treatment of Progranulin Insufficiency From GRN Gene Mutations
Brief Title: Dose Finding Study of Nimodipine for the Treatment of Progranulin Insufficiency From GRN Gene Mutations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: The Bluefield Project to Cure Frontotemporal Dementia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CHR12-09098
Record Dates: First submitted 2013-03-27; First posted 2013-04-19 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-05

CONDITIONS: Progranulin Mutation Carriers
MeSH Terms: interventions — Nimodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nimodipine (Experimental)
  Interventions: Drug: Nimodipine

INTERVENTIONS:
Drug: Nimodipine — Nimodipine is an FDA-approved drug for subarachnoid hemorrhage indication
  Other Names: Nimotop

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose of nimodipine as well as the safety and tolerability of oral nimodipine in progranulin mutation carriers in preparation for longer term efficacy studies in patients with frontotemporal dementia due to progranulin gene mutations.

DETAILED DESCRIPTION:
8 people with a GRN gene mutation will be given escalating doses of oral nimodipine for four weeks, followed by the maximally tolerated dose for four weeks. To maximize enrollment, the trial will enroll both symptomatic and asymptomatic GRN mutation carriers. The trial will include a four week, dose-escalation phase followed by 1-month maintenance phase, and a 1-week taper. Assessments at the study site will take place prior to starting nimodipine, each week the dose is increased (weeks 1-5), after 4 weeks of maintenance dose, and 2 weeks after completion of the study. These will include blood chemistry tests, ECGs, and blood pressure. Both dose escalation and maintenance will focus on safety and tolerability of nimodipine treatment in this population as well as plasma progranulin levels as a biomarker outcome. The trial will incorporate a variety of other fluid biomarker (blood and CSF) and imaging assessments to determine which will be most sensitive to nimodipine pharmacodynamic effects in this population.

ELIGIBILITY:
Inclusion Criteria (all must be met):

* Signed and dated written informed consent obtained from the subject and/or the subject's caregiver in accordance with local IRB regulations
* Symptomatic GRN mutation carrier as defined by presence of known disease-associated GRN mutation confirmed by genetic testing and meeting international (2011) criteria for FTD (Rascovsky et al., 2011), Boeve (2003) criteria (B. F. Boeve, Lang, & Litvan, 2003) for CBS, or Gorno-Tempini criteria (2011) for primary progressive aphasia (Gorno-Tempini et al., 2011) (gene carrier status known) OR
* Asymptomatic GRN mutation carrier (gene carrier status known) from family with known disease-associated mutation;
* Age: >30
* MMSE ≥ 10 at screening visit.
* Judged by investigator to be able to comply with all study procedures
* In the opinion of the investigator, the patient will be compliant with the protocol and have a high probability of completing the study
* Lack of other recent, severe medical conditions.

Exclusion Criteria(Any one of the following will exclude a subject from being enrolled into the study):

* Hypersensitivity or other contra-indication to nimodipine use
* Systemic autoimmune disease (such as rheumatoid arthritis, thyroid disease, or diabetes) that might alter progranulin levels.
* Regular use of systemic corticosteroids or other anti-inflammatory medication. NSAID use acceptable if on a stable dose for 30 days prior to screening and agrees to remain on same dose for duration of trial.
* Subject is pregnant, plans to become pregnant during course of study or has a positive urine pregnancy test.
* Unwilling to use two forms of contraception if not surgically sterile for duration of study.
* History of cancer (other than basal cell CA of skin) within 5 years.
* History of myocardial infarction, cardiac conduction block, arrhythmia or other significant cardiac illness in the opinion of the investigator (in consultation with a board certified cardiologist).
* History of peptic ulcer.
* Metabolic disease such as gout or poorly controlled diabetes.
* History of alcohol or substance abuse within 1 year prior to screening, if deemed clinically significant by investigator.
* Any current malignancy, or any clinically significant hematological, endocrine, cardiovascular, renal, hepatic, gastrointestinal or neurological disease. If the condition has been stable for at least the past year and is judged by the investigator not to interfere with the patient's participation in the study, the patient may be included.
* CT or MRI evidence of any of the following: hydrocephalus, stroke, space-occupying lesion, cerebral infection or any clinically significant CNS disease other than FTD, CBS, or progressive aphasia.
* Systolic blood pressure greater than 180 or less than 90 mm Hg. Diastolic blood pressure greater than 105 or less than 50 mm Hg.
* Abnormal ECG at screening and judged to be clinically significant by the investigator and/or board certified cardiologist.
* Use of investigational drugs or participation in investigational drug study within 30 days of screening or 5 half lives of the previous investigational drug, whichever is longer.
* Use of nimodipine within the 4 weeks prior to start of trial.
* Within 4 weeks of beginning or during the course of the study, concurrent treatment with calcium channel antagonists, blood thinners (e.g. clopidogrel, warfarin), or statin medication in combination with niacin.
* Clinically significant lab abnormalities at screening, including creatinine ≥ 1.7, B12 below laboratory normal reference range, or TSH above site's laboratory normal reference range. Subjects with abnormal B12 or TSH levels at screening may be included per investigator's discretion.
* Contraindication to MRI examination for any reason (e.g., severe claustrophobia, ferromagnetic metal in body).

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-03; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Maximum dose tolerated of nimodipine | up to 10 weeks
  Nimodipine dose will be increased weekly for four weeks then maintained for 4 weeks at highest tolerated dose, followed by a 1-week taper.

SECONDARY OUTCOMES:
Plasma progranulin levels | up to 10 weeks post initial dosing
  Plasma progranulin levels will be obtained at screening, baseline, and at each week dose is increased, after the 4 week maintenance phase, and 2 weeks after the taper. Due to the small sample size, inferential statistics will not be calculated to assess the endpoints of interest. However, descriptive statistics will be presented for the primary and secondary outcome measures (such as plasma and CSF progranulin levels) summarized by treatment group and visit. For these continuous variables, the following information will be presented by visit: n, mean, standard deviation and order statistics (minimum, 25th percentile, median, 75th percentile and maximum). These statistics will be presented using the actual value at baseline and the change from baseline for later data.
Inflammatory marker levels (ESR, CRP, cytokines) | up to 10 weeks post initial dosing
  Markers of inflammation will be obtained from the blood at screening, baseline, each week dose is increased, after 4 weeks of stable dose, and 2 weeks after the taper. Due to the small sample size, inferential statistics will not be calculated to assess the endpoints of interest. However, descriptive statistics will be presented for the primary and secondary outcome measures (such as plasma and CSF progranulin levels) summarized by treatment group and visit. For these continuous variables, the following information will be presented by visit: n, mean, standard deviation and order statistics (minimum, 25th percentile, median, 75th percentile and maximum). These statistics will be presented using the actual value at baseline and the change from baseline for later data.
CSF progranulin | baseline (week 1) and 8 weeks after initial dosing
  CSF progranulin levels will be obtained at baseline and week 8
CSF cytokines | baseline (week 1) and 8 weeks post dosing
  CSF cytokines will be obtained at baseline and after 8 weeks of taking nimodipine
Brain MRI scan | Screening and week 8
  To acquire preliminary data on the sensitivity of functional and brain MR imaging (resting-state functional connectivity and arterial spin label perfusion) to progranulin elevating therapies.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Boxer, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Memory and Aging Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data analysis is underway